CLINICAL TRIAL: NCT03846440
Title: Inadequate Protein Intake at Specific Meals and Functionality in Middle to Older Aged Mexican Adults
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Hospital General de Occidente (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Sport, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: HGO-ICAAFYD18-2
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Aging
Keywords: Protein intake; Older adults; Mexican adults; Functionality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Middle to older aged (>50 years) Mexican adults attending to the Geriatrics Department from the Western General Hospital (Zapopan, Jalisco,Mexico).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
This study sought to determine if the inadequate protein intake per meal (defined as eating <30 g protein or 0.4 g protein/kg body mass) at specific meals (breakfast, lunch, dinner) is associated with functionality in middle to older aged Mexican adults. Functionality was evaluated with self-reported questionnaires to assess their functionality score for different activities of daily living.

DETAILED DESCRIPTION:
Detailed dietary information was obtained for each participant to estimate dietary protein intake per meal (breakfast, lunch, dinner). One meal was considered with inadequate protein intake if its content was <30 g or 0.4 g/kg.

Functionality was assessed with two validated questionnaires. One for instrumental activities of daily living (Lawton) and another for activities of daily living (Barthel). We calculated a score according to each author's scales. This score was divided into three possible groups as "low", "middle", and "high" scores.

To analyze the association between inadequate protein intake per meal and functionality, we used multinomial logistic regression. The outcome variable was functionality ("High" was the reference group, "middle" and "low" scores were considered as impaired functionality), and the predictive variables were inadequate protein intake at breakfast, lunch, and dinner. They were adjusted for age, BMI categories, number of diagnosed diseases, sex, and inadequate protein intake per day (<1.2 g/kg/d).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to stand up and walk independently or with walking sticks only.
* Subjects able to answer questionnaires independently or with minimum caregivers' assistance.

Exclusion Criteria:

* Subjects reporting any kind of hospitalization within the last year.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle to older aged Mexican adults attending to the Geriatrics Department at the Western General Hospital (Hospital General de Occidente) for their usual medical screening or first time assessment.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Functionality on Instrumental Activities of Daily Living | One day
  Functionality score for instrumental activities of daily living (assessed with Lawton questionnaire). This instrument assess how well the subject perform some daily activities involving tools (e.g. handling finances, taking medication, using the telephone). The instrument consists on five items for men and eight for women, and each item is coded for 0 or 1 depending on if subjects are capable to successfully complete the activity. Therefore, the score ranges from 0 to 5 in men and 0 to 8 in women, the higher the score, the more functional the subject.
Functionality on Activities of Daily Living | One day
  Functionality score for activities of daily living (assessed with Barthel questionnaire). This instrument assess how well the subject perform some daily activities (e.g. dressing, using stairs). The instrument consists on ten items for both men and women coded as 0 or multiples of 5 (i.e. 5, 10, 15) depending on if subjects are capable to successfully complete the activity. The score ranges from 0 to 100 for both men and women, the higher the score, the more functional the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gaytán-González, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided